CLINICAL TRIAL: NCT02797483
Title: Multi-country Studies on the Effect of Positional Distribution of Fatty Acids at the Triglyceride Backbone of Vegetable Oils on Fat Deposition and Selected Health Outcome Measures - Malaysia
Brief Title: Multi-country Study- Effect of Dietary Fats on Fat Deposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: IMU University, Malaysia (Other); Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PD 205/15 (b)
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Fat Blue (Experimental): 16 weeks interventions
  Interventions: Other: Test Fat Blue
- Test Fat Green (Experimental): 16 weeks interventions
  Interventions: Other: Test Fat Green
- Test Fat Red (Experimental): 16 weeks interventions
  Interventions: Other: Test Fat Red

INTERVENTIONS:
Other: Test Fat Blue — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment Test Fat Blue which incorporated into daily snacks (~50g of test fats, 2 experimental cupcakes (~15g test fat each) for breakfast and 4 pieces experimental cookies (~5g test fat each) for afternoon tea together with a palm olein-based background diet for 16 weeks.
  Arms: Test Fat Blue
Other: Test Fat Green — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment Test Fat Green which incorporated into daily snacks (~50g of test fats, 2 experimental cupcakes (~15g test fat each) for breakfast and 4 pieces experimental cookies (~5g test fat each) for afternoon tea together with a palm olein-based background diet for 16 weeks.
  Arms: Test Fat Green
Other: Test Fat Red — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment Test Fat Red which incorporated into daily snacks (~50g of test fats, 2 experimental cupcakes (~15g test fat each) for breakfast and 4 pieces experimental cookies (~5g test fat each) for afternoon tea together with a palm olein-based background diet for 16 weeks.
  Arms: Test Fat Red

SUMMARY:
There is existing evidence to show that vegetable oils having unsaturated fatty acids in the sn-2 position with predominantly palmitic acid (C16:0) or stearic acid (C18:0) in the sn-1 and sn-3 positions of fat molecules do not raise serum cholesterol levels. These observations have come to be known as or explained by the "sn-2 hypothesis". New evidence have also emerged to show that saturated fatty acids (C16:0, C18:0) in the sn-1 and -3 positions reduces fat deposition in a rat model. Therefore, further studies in humans are warranted to confirm these earlier findings.

Fats and oils are made up of >90% triacylglycerol (TAG)- fat molecules which consist of a glycerol backbone to which 3 esterified fatty acids are attached. The positions of fatty acid attachment are referred to by stereospecific numbers, sn -1, -2 and -3. Early evidence shown that the unique stereospecificity of fatty acid distribution on the palm fat molecule conferred health benefits in that it inhibited experimental atherosclerosis in the rabbit model.

In vegetable oils, oleic acid [a monounsaturated fatty acid (MUFA)] is predominantly situated at the sn-2 position, while in animals fats it is predominantly palmitic acid or stearic acid (C16:0 or C18:0-saturated fat) that is situated there. Even though palm olein and lard have similar proportions of saturated fatty acid (SFA), MUFA and polyunsatuared fatty acid (PUFA), they differ significantly in their positional distribution on the TAG molecule. Palm olein TAG contains only 7-11 % palmitic acid at the sn-2 position while about 87% is unsaturated fatty acids (oleic acid and linoleic acid). Lard has the highest amount of palmitic acid in the sn-2 position at 70%. On the other hand, in human milk, palmitic acid is predominantly in sn-2 (53-57 %) while cow milk fat contains less palmitic acid (38 %) there. It is now believed that the distribution of fatty acids in the TAG is more important than the fatty acid composition alone in conferring the oils' 'saturated' or 'unsaturated' properties.

In this proposed study, the effects on the outcome measures investigated of different fatty acids (palmitic acid, oleic acid, linoleic acid) at the sn-1, sn-2 and sn-3 positions of the TAG molecule in three different test fats will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female, aged 20-60 years
* BMI 18-5-27.5 kg/m2

Exclusion Criteria:

* History of any one of these chronic diseases - type 2 DM, hypertension, coronary heart disease, hyperlipidemia, liver disease, cancer
* Current problem with indigestion or constipation or bowel movement
* On medication/nutraceutiucals to reduce blood lipids or blood pressure or weight
* Pregnant or lactating women or taking COCP
* Habitual smokers (>2 sticks per day)
* Alcoholism (>21 units per week for men & >14 units per week for women)
* Mean screening blood pressure >140/90 mmHg
* Screening TC>6.2 mmol/L or TAG >2.0 mmol/L
* Planned trip abroad/overseas during period of study
* Unable to adhere to at least 90% of the prescribed oil & recommended energy and fat per day per research protocol

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of liver fat content | week 0 (baseline) and week 16
  measured by magnetic resonance imaging (MRI) scan

SECONDARY OUTCOMES:
Change of body mass index (BMI) | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Tanita Segmental Body Fat Analysis
Change of waist circumference | week 0 (baseline), week 4, week 8, week 12 and week 16
Change of body fat distribution/content | week 0 (baseline), week 4, week 8, week 12 and week 16
Change of visceral adiposity index (VAI) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by visceral adiposity index (VAI)
Change of body adiposity index (BAI) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by visceral body adiposity index (BAI)
Change of serum leptin | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by enzyme-linked immunosorbent assay (ELISA) development kits
Change of serum total cholesterol (TC) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
Change of serum high-density lipoprotein cholesterol (HDLC) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
Change of serum triacylglycerie (TAG) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
Change of serum low-density lipoprotein (LDLC) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
Change of serum lipoprotein ration (TC/HDLC) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
Change of serum HDL-subfractions | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Lipoprint® HDL Subfractions Test
Change of serum LDL-subfractions | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Lipoprint® LDL Subfractions Test
Change of serum Apolipoprotein A | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Siemens Advia 2400 Chemistry Analyzer
Change of serum Apolipoprotein B | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Siemens Advia 2400 Chemistry Analyzer
Change of serum Lp (a) | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by Siemens Advia 2400 Chemistry Analyzer
Faecal fatty acid composition (FAC) | week 0 (baseline), week 4, week 8, week 12 and week 16
  FAC of faecal extracted fat measured by gas chromatography (GC)
Change of visceral adipose tissue | week 0 (baseline) and week 16
  measured by MRI
Change of subcutaneous adipose tissue | week 0 (baseline) and week 16
  measured by MRI
Change of serum interleukin-6 (IL-6) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by ELISA development kits
Change of serum tumor necrosis factor alpha (TNF-α) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by ELISA development kits
Change of serum high-sensitivity C-reactive protein (hsCRP) | week 0 (baseline), week 4, week 8, week 12 and week 16
  analysed by ELISA development kits
Systolic and diastolic blood pressure | week 0 (baseline), week 4, week 8, week 12 and week 16
  measured by blood pressure meter

CONTACTS AND LOCATIONS:
Overall Officials: Choo Yuen May, PhD, Study Chair — MPOB; Augustine Ong Soon Hock, PhD, Principal Investigator — MPOB; Voon Phooi Tee, PhD, Principal Investigator — MPOB; Tony Ng Kock Wai, PhD, Principal Investigator — IMU; Verna Lee Kar Man, PhD, Principal Investigator — IMU; Norhaizan Mohd Esa, PhD, Principal Investigator — UPM; Teh Soek Sin, PhD, Principal Investigator — MPOB; Yap Sia Yen, PhD, Principal Investigator — MPOB; Ng Yen Teng, Bsc, Principal Investigator — MPOB

IPD SHARING:
Plan to Share IPD: Undecided